CLINICAL TRIAL: NCT06444412
Title: GA-68 PSMA-11 PET To Evaluate Malignant Glioma Recurrence - A Pilot Study
Brief Title: An Investigational Scan (Ga-68 PSMA-11 PET/CT) for Detection of Disease Recurrence or Progression in Patients With Glioma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CR250101; NCI-2024-03913 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-007985 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-05-31; First posted 2024-06-05 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: WHO Grade 3 Glioma; WHO Grade 4 Glioma
MeSH Terms: interventions — gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (Ga-68 PSMA-11, PET/CT) (Experimental): Patients receive Ga-68 PSMA-11 IV and then undergo PET/CT over 1 hour, 50-100 minutes after injection.
  Interventions: Procedure: Computed Tomography; Other: Electronic Health Record Review; Drug: Ga 68 PSMA-11; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Other: Electronic Health Record Review — Ancillary studies
Drug: Ga 68 PSMA-11 — Contrast dye given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; AAA 517; AAA-517; AAA517; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; Ga 68 PSMA-11, Intravenous Solution; Gallium Ga 68 PSMA-11; Gallium Ga 68-labeled PSMA-11; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This clinical trial evaluates whether gallium-68 (Ga-68) prostate specific membrane antigen (PSMA)-11 positron emission tomography (PET)/computed tomography (CT) imaging is useful in differentiating between disease that has come back after a period of improvement (recurrence) or that is growing, spreading, or getting worse (progression) and treatment effect in patients with glioma. Patients with glioma undergo frequent imaging for assessment of disease status. After first-line treatment however, the correlation between imaging findings and tumor activity can be confused, and surgery is often required for definitive diagnosis. The PET/CT scanner is an imaging machine that combines 2 types of imaging in a single scan. The PET scanner detects and takes pictures of where the radioactive imaging agent (68Ga PSMA-11) has gone in the body and the CT scanner uses x-rays to take structural pictures inside the body. PSMA PET also binds to neoplastic blood vessels, including those in gliomas. This study may help researchers learn whether GA-68 PSMA-11 PET/CT is useful for improving detection of tumor recurrence or progression, as opposed to treatment effects, in patients with gliomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the feasibility and immediate safety profile of gallium Ga 68 gozetotide (Ga-68 labeled PSMA-11) brain PET in patients with gliomas, assessed as the percentage of patients who experience grade 3 or higher adverse effects deemed to be at least possibly related to PSMA-11 occurring prior to the patient leaving the Nuclear Medicine department.

EXPLORATORY OBJECTIVES:

I. An exploratory investigation will be performed in regions of high tumor cell density (tumor recurrence) and low tumor cell density/treatment effect to determine whether PSMA-11 uptake differs significantly between true tumor progression vs. in radiation treatment effects by performing a radiology-pathology comparison of visual and descriptive features of the PET with biopsy.

II. To identify optimal maximum standardized uptake value (SUVmax) thresholds for differentiating viable tumor from treatment effect.

III. To perform a radiology-pathology correlation of PSMA uptake at PET with tumor PSMA immunohistochemistry (IHC) immunostaining, tumor pathology features, and signal and enhancement characteristics at magnetic resonance imaging (MRI) (no research MRI will be obtained, based on MRI images obtained for clinical use).

IV. To evaluate the added diagnostic value of Ga-68 PSMA-11 PET beyond MRI (using information from a clinical MRI[s] obtained prior to enrollment in the study) for detecting viable enhancing tumor from treatment effects.

OUTLINE:

Patients receive Ga-68 PSMA-11 intravenously (IV) and then undergo PET/CT over 1 hour, 50-100 minutes after injection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* History of World Health Organization (WHO) grade III or IV infiltrating glioma previously treated with first-line chemoradiotherapy.
* MRI findings compatible with contrast-enhancing recurrent infiltrating glioma.
* Planned craniotomy for resection of suspected disease recurrence.
* Willing to sign release of information for any radiation and/or follow-up records.
* Ability to provide informed written consent.
* Ability to provide tissue for mandatory correlative research component.

Exclusion Criteria:

* Unable to undergo a PSMA PET/CT scan (e.g. body habitus, claustrophobia).
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential unwilling to employ adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (safety and tolerability) | Up to 24 hours after 68Ga-PSMA-11 injection
  Assessed as the percentage of patients who experience Grade 3 or higher adverse effects deemed to be at least possibly related to PSMA-11. Adverse effects will be assessed according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.
Tolerability of PSMA positron emission tomography scan | Up to 60 days
  Will assess any issues in completion of the PSMA positron emission tomography scans in these patients and summarize those in a descriptive manner.

CONTACTS AND LOCATIONS:
Overall Officials: Brian J. Burkett, MD, MPH, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials